CLINICAL TRIAL: NCT00620880
Title: Performance of CAST With Different Allergens in Patients With Cat Dander Allergy
Brief Title: IVN-CAT-001A Performance of CAST With Different Allergens in Patients With Cat Dander Allergy
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: ImVision AG (Unknown)
Responsible Party: University Hospital Zürich, University of Zurich
Other Study IDs: IVN-CAT-001A
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Allergy to Cats
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Blood sample

SUMMARY:
Primary objective of the trial:

To determine at which concentration the fusion protein MAT Fel d1 degranulates basophils of cat dander allergic patients, in comparison to a cat dander extract and to Fel d1 alone

ELIGIBILITY:
Inclusion criteria: 1. Patient with Cat Dander Allergy evidenced by positive history 2. Age: 18 to 75 years

Exclusion criteria: 1. Use of oral corticosteroids, Chromoglycin, Ketotifen, or any immunosuppressive drugs within the last 2 months 2. Psychiatric disorder resulting in malcompliance 3. Neg. IgE to Cat dander

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland